CLINICAL TRIAL: NCT03671616
Title: Immunogenicity and Safety of Adjuvanted Reduced Dose Inactivated Polio Vaccine, IPV-Al SSI Given as a Booster Vaccination at the Age of 15-18 Months to Infants Previously Immunised With IPV-Al SSI or IPV SSI
Brief Title: Immunogenicity and Safety of Adjuvanted Reduced Dose Inactivated Polio Vaccine Given as a Booster at Age 15-18 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Larix A/S (Industry); Vaxtrials S.A. (Other); AJ Vaccines A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VIPV-07 E1
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPV-Al SSI (Experimental): Single arm trial. All subjects will receive the IPV-Al SSI as booster vaccination
  Interventions: Biological: IPV-Al SSI

INTERVENTIONS:
Biological: IPV-Al SSI — IPV-Al contains the reduced dose of IPV to be administered intramuscularly to the anterolateral of the right thigh. A single dose of the IPV-Al SSI will be given to infants age 15-18 months.

SUMMARY:
This is a phase III assessing the safety and immunogenicity of adjuvanted the reduced dose inactivated polio vaccine, IPV-Al SSI given as a booster vaccination to infants who were previously immunised with primary vaccination of IPV-Al SSI or IPV SSI in the VIPV-07 trial at age 2, 4, and 6 months. The IPV-Al SSI vaccine will be given at the age of 15-18 months.

DETAILED DESCRIPTION:
At Visit 1 (screening, blood sample, and vaccination), the subject's eligibility is assessed according to the pre-specified in-/exclusion criteria. Information on medical history, and concomitant medication are collected and a physical examination is performed and vital signs are measured (demographics data is captured from the VIPV-07 database). The health assessment of the subject will include measurement of height, weight, temperature, heart rate, respiratory rate (breathing) and a general physical examination (which can include skin, head, eyes, ears, nose, throat, heart, lungs, lymph nodes, abdomen, and the musculoskeletal system). A pre-vaccination blood sample is taken for polio antibody determinations. The subject is vaccinated with IPV-Al (and concomitant vaccine(s) according to national guidelines, if relevant) and subsequently observed for immediate adverse events 30 minutes after the vaccination. An eDiary, a thermometer and a ruler are handed out to the parent(s)/guardian(s) for measurements and recording of temperature, injection site reactions and solicited systemic adverse events (AEs). These activities are performed daily, starting on the day of the vaccination and the following 2 days and until resolved. Any other AEs are recorded in the eDiary as instructed by the trial staff. A contact to the parent(s)/guardian(s) via telephone will be made after the vaccination visit to remind and check if the parent(s)/guardian(s) have any questions regarding how to fill in the eDiary.

At Visit 2 (blood sample and trial completion), 1 month after Visit 1, the eDiary is collected, adverse events and concomitant medications are recorded, a blood sample for poliovirus antibody determination is taken and the end of the trial page is completed.

In addition to the trial vaccine, the trial subjects will receive concomitant routine childhood vaccinations. The trial vaccine is administered in the anterolateral aspect of the right thigh, whereas the other injectable childhood vaccines are administered in the left thigh.

ELIGIBILITY:
Inclusion Criteria:

1. Infants having completed the VIPV-07 trial
2. Healthy assessed from medical history and physical examination
3. Parent(s)/guardian(s), according to the local legal requirements, have been properly informed about the trial and have signed the informed consent form
4. Parent(s)/guardian(s), according to the local legal requirements, have granted access to the infant's trial related medical records
5. Parent(s)/guardian(s), according to the local legal requirements, are likely to comply with trial procedures

Exclusion Criteria:

1. Previously vaccinated with OPV
2. Previously vaccinated with IPV outside the VIPV-07 trial
3. Known or suspected immunodeficiency (e.g. leukaemia or lymphoma) or family history of congenital or hereditary immunodeficiency. HIV infection is not an exclusion criterion
4. Severe uncontrolled chronic disease (e.g. neurologic, pulmonary, gastrointestinal, hepatic, renal or endocrine)
5. Known or suspected allergy to vaccine constituents (e.g. hypersensitivity to formaldehyde, aluminium or 2-phenoxyethanol)
6. Previous Yellow Fever vaccination
7. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections or blood sampling
8. In treatment with systemic corticosteroids given p.o., i.v., i.m. ≤ 1 month prior to inclusion or during the trial. Subjects administered corticosteroid topically or by asthma inhalators are eligible for inclusion
9. Treatment with a product, which is likely to modify the immune response (e.g blood products and immunoglobulins) ≤ 3 months prior to inclusion or planned during the trial period
10. Participating in another interventional clinical trial
11. Not suitable for inclusion in the opinion of the investigator

Ages: 15 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 666 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Booster effect ratiors of GMT | Change from Visit 1 (6-9 months post-3rd vaccination) to one month after booster vaccination (Visit 2)
  Booster effect (day 28 / day 0 titres), from individual serum titre values for antibodies against poliovirus types 1, 2 and 3 measured before and one month after the booster vaccination

SECONDARY OUTCOMES:
Seroprotection rates before booster vaccination | 6-9 months post-3rd vaccination
  Subjects with seroprotection (titre ≥ 8) against poliovirus types 1, 2 and 3 before the booster vaccination.
Seroprotection rates after booster vaccination | one month after booster vaccination
  Subjects with seroprotection (titre ≥ 8) against poliovirus types 1, 2 and 3 one month after the booster vaccination.
GMT value before booster vaccination | 6-9 months post-3rd vaccination
  Geometric mean antibody titres (GMTs) against poliovirus types 1, 2 and 3 before the booster vaccination.
GMT value after booster vaccination | one month after booster vaccination
  GMTs against poliovirus types 1, 2 and 3 one month after the booster vaccination.
Number of adverse events | 6-9 months post-3rd vaccination and one month after booster vaccination
  All adverse event
Persistence (tite rates) of antibodies | 6-9 months post-3rd vaccination and one month after booster vaccination
  Persistence of antibodies against poliovirus types 1, 2 and 3 in subjects previously im-munised with IPV-Al SSI or IPV SSI

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Kromann, Study Director — Statens Serum Institut
Locations (1):
- Cevaxin, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes
EudraCT
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Saez-Llorens X, Thierry-Carstensen B, Stoey LS, Sorensen C, Wachmann H, Bandyopadhyay AS, Nielsen PI, Kusk MV. Immunogenicity and safety of an adjuvanted inactivated polio vaccine, IPV-Al, following vaccination in children at 2, 4, 6 and at 15-18 months. Vaccine. 2020 May 6;38(21):3780-3789. doi: 10.1016/j.vaccine.2020.02.066. Epub 2020 Apr 6. PMID 32273184